CLINICAL TRIAL: NCT06107244
Title: A Mixed Methods Investigation of Paramedic Independent Prescribing in Emergency and Urgent Care.
Brief Title: Paramedic Independent Prescribing in Emergency and Urgent Care
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS Number: 310457
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Prescribing; Prescribing Practices; Prescribing Tendencies; Prescribing Decisions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this mixed methods observational study is to investigate paramedic independent prescribing (PIP) in emergency and urgent healthcare settings.

The main questions it aims to answer are:

1. What are benefits and limitations of paramedic independent prescribing in emergency and urgent care settings and how does it contribute to patient care and healthcare service delivery?
2. What facilitators and barriers exist which influence the implementation and delivery of PIP as a new and complex intervention within emergency and urgent care?

Participants in the study will include paramedics qualified in PIP and staff working at the case study sites. With participant consent, data will be collected using non-participant observation of the prescribing practice of 4-6 paramedics at each site, capturing this data through field notes. The views and insights of a range of other site staff such as managers, doctors and other clinicians will be interviewed at each case site, during semi structured interviews.

At each case site anonymised prescribing frequency data will also be collected to understand the range and frequencies of prescribed medication by paramedics. Relevant meetings (such as clinical governance and medicines management meetings) will also be observed, and documentary analysis of relevant site documents will also be undertaken.

DETAILED DESCRIPTION:
This research study aims to investigate paramedic independent prescribing (PIP) within emergency and urgent healthcare, whilst also exploring any facilitators or barriers to its implementation and delivery. NHS emergency and urgent care is currently facing an unprecedented level of demand. Advanced level paramedics are able to help meet the challenges faced, by providing autonomous high-level care both in ambulance services, within the emergency departments (EDs) and in urgent care services.

Since 2018, advanced paramedics have been able adopt PIP and it is anticipated that this will enhance their ability to independently provide patient care in a range of settings. However, very little previous research has been undertaken to evaluate PIP. It is therefore unclear if and how PIP is benefiting patients and NHS services, or if any improvements are required to maximise its potential. Several potential issues may also exist, which include an inability to prescribe certain medicines known as controlled drugs (which include pain medication and sedatives), variation in the training and education of prescribing, alongside concerns about organisational readiness and support for PIP in ambulance services.

The research detailed here is the final element of a larger mixed methods Doctoral research project. Previous work has included a systematic literature review conducted in 2021-2022 which focused on synthesising the findings of the very limited amount of research on PIP and the larger body of research evidence on independent prescribing by other healthcare professionals working in emergency and urgent care settings. Semi structured interviews were also conducted with PIP key stakeholders and subject experts (n=15) between October 2022-January 2023, to explore their higher level views on PIP. Participants included senior NHS leaders and directors from a range of settings where PIP is utilised. These including ambulance Trusts and emergency departments and urgent care services. Participants also included higher education leaders involved with the delivery of PIP education, and national leaders from Health Education England and the College of Paramedics.

In order to answer the research question and aims as part of a convergent mixed methods design, case study research will now be conducted in two different emergency and urgent care settings where paramedics utilise PIP. These will include paramedic advanced clinical practitioners in emergency medicine (ACP-EM) within an ED setting and paramedic practitioners in an integrated urgent care service.

Over the 6-8 month data collection period, a range of data will be collected. These will include quantitative data in the form of prescribing frequency data for all prescribing paramedics employed at each site, non-participant observation of of prescribing practice by paramedics at each site, semi-structured case study interviews with a range of site staff, documentary analysis of relevant documents and observation of relevant meetings or events.

Non-Participant Observation and Informal Reflective Conversations:

A total of 4-6 prescribing paramedics will be recruited in each case study site and observed using non-participant observation. This is anticipated to occur during 4-6 10 hour shifts per participant. Observations and field notes will be focused on collecting data regarding any prescribing activity undertaken.

During these shifts, informal reflective conversations will also be held with each recruited paramedic at appropriate times, to discuss and probe emerging issues around the prescribing activity observed, or to ask questions about this. These conversations will also be used to discuss the research aims with participants in a naturalistic manner and gain their views and perceptions around these.

Brief field notes (or jottings) will be initially made whilst in the field, using Microsoft OneNote on an Apple iPad Pro, and will then be expanded on after the shift oOnce written, full field note data will be stored, managed and analysed within NVivo computer software.

Review of prescribing data and relevant site documentation:

With the assistance of research staff and local collaborators at each site, the researcher will obtain and review anonymised prescribing frequency data for all prescribing paramedics at each site from the previous 12 months. Frequency data will be analysed using SPSS to generate descriptive statistics.

Relevant site documentation will also be requested for review, such as independent prescribing policies, prescribing paramedic job descriptions and role specifications, internal prescribing formularies and organisational guidance for paramedic prescribers at the site. All relevant documents will be imported into NVivo and will be coded and categorised alongside the field note data.

Case Study Interviews:

Semi structured, case-study interviews will also be undertaken with a range of staff at each case site, to explore their views and perceptions regarding PIP. Following scoping work and engagement with potential sites, it is anticipated that between 10-15 interviews will be conducted per site during the 6-8 month data collection period. Engagement work with site staff and expert advisors from the College of Paramedics Medicines and Prescribing Special Interest Group was undertaken to discuss the potential range of interview participants. These will therefore include senior and junior grade doctors, independent prescribing leads within the organisation, clinical managers, clinical directors and other healthcare professionals at the site, including nurses and non-prescribing paramedics.

Whilst this engagement work has been used as part of the research design process, additional work will be undertaken when in the field to identify potential participants, by seeking recommendations from the recruited prescribing paramedics and from any recruited interview participants. Any potential participants identified by the recruited prescribing paramedics or interview participants, will be contacted by local collaborators such as clinical and research managers through their organisational email address. Local site collaborators or research staff will be asked to send an introductory email to them, which will contain a participant information sheet and consent form. Potential interview participants will be asked to sign and return the consent form to the researcher by email should they wish to participate. Up to two reminder emails will be sent to potential participants by local collaborators, at two week intervals. Any staff who decline to participate will not be sent further reminder emails.

It is anticipated that interviews will last 15-30 minutes and will be conducted when staff are not directly engaged in patient care. This may include during rest breaks, in-between patient cases or during administration time. Interviews will either be conducted face to face whilst on site, or using video conferencing such as Microsoft Teams, to engage with staff flexibly. This will include being able to interview participants who are not on site when it is convenient to speak with them. Permission will be sought from participants to audio record the interviews, to facilitate transcription and analysis. The recordings will then be deleted once this process has been completed. Both for face to face and online interviews, audio recordings will be captured on an iPad Pro. Audio data will be synced and stored on a secure University OneDrive Account and not locally on the device. Furthermore, the device is secured with a complex password and Face ID technology. Only the researcher will have access to this device, both in the field and when it is not in use and stored and their home address.

Interviews will be guided by an interview topic guide, framed around the research question and objectives. However the interview will be participant led, given the focus and content will likely vary, depending on the specific role of participants. For example, interviews with doctors might focus more on medical support for PIP, whilst interviews with site managers may focus on organisational support for PIP. The interview topic guide has been informed by the topic guide and interview data from the key stakeholder interviews previously undertaken.

Meeting Observations:

Opportunities to observe relevant meetings will also be sought during the data collection period. For example, medicines governance/management meetings. It is also anticipated some of these meetings may be held online. The approach to data collection during these meetings will be the same as for the non-participant observations, recording brief notes or jottings which will be expanded through more detailed field notes following the meeting. In order to facilitate this process, the researcher will request to audio record the meeting. If permitted to do so, the audio recordings will then be deleted once the detailed field notes have been written, again with the assistance of auto transcription software, combined with accuracy checks by the researcher.

Data Analysis:

The full field notes from observations of and informal conversations with prescribing paramedics, observed meetings and case study interviews transcripts, alongside relevant extracts from site documents will be used to triangulate data from all sources and to produce a detailed or "thick description" of the research setting and its participants. Field note data will be used to support ongoing assessment by the researcher and their supervisory team, to ensure data saturation has been achieved in each case. If required, additional observations shifts will be negotiated with participants,

Data from these sources will be coded and categorised within NVivo computer software, to facilitate a process of concept mapping, which will examine if and how each item of data coded belongs to a particular category, noting its similarities with and differences from other data categorized, including data from other case study sites. Coding and categorisation of the data in this way will facilitate an inductive approach to generating themes or typologies. NVivo software will be used to store and manage this research data and will facilitate the data analysis process of coding, categorisation, concept mapping, and the generation of themes or typologies across the dataset. All research data will be anonymised before transferring to Nvivo and participants will be assigned a unique identifier (participant number and basic details of their role eg prescribing paramedic-1).

Triangulation of data within each site will be undertaken, whereby data from the guided conversation case-study interviews, nonparticipant observation, meeting observations, documentary analysis and prescribing records are analysed and compared to develop converging lines of enquiry. Cross case analysis of case study sites will also be undertaken, to assess if and how the data from each case replicates or contrasts each other. Case study data analysis will be produced using both a narrative form and using matrices- whereby data is placed into a visual matrix of categories to facilitate analysis and the identification of patterns, insights or concepts.

As part of a convergent mixed methods design, the quantitative case study data, in the form of prescribing frequency statistics and the qualitative data from field notes will be integrated through narrative analysis, joint displays and using matrices, to facilitate integration of the case study data with the previous research work packages of a critical narrative review and key stakeholder interviews. NVivo software will be used to store and manage all research data during the study and to facilitate the data analysis process.

Adam Bedson, Clinical Doctoral Research Fellow, (NIHR302127) is funded by Health Education England (HEE) / National Institute for Health Research (NIHR) for this research project. The views expressed in any related publications/outputs are those of the authors and not necessarily those of the NIHR, NHS or the UK Department of Health and Social Care.

ELIGIBILITY:
Inclusion Criteria for Paramedic Prescriber Participants:

* Registered Paramedic
* Completion of an approved IP course and annotated as a PIP with the Health Care Professions Council
* Registered as an independent prescriber with employing Trust and using PIP in emergency and urgent care practice.
* Working in a role which is focused on the assessment of emergency and urgent care presentations. This includes undifferentiated minor and major illness and injury, urgent palliative care cases during out of hours periods and medical emergencies.

Exclusion Criteria for Paramedic Prescribing Participants:

* Paramedics who are not qualified or registered in IP, including those currently undertaking their training
* Paramedics qualified in PIP but not actually independently prescribing in practice
* Prescribing paramedics working in roles that are not associated with emergency and urgent care. This includes pre hospital critical care paramedic roles and those working in areas of secondary care outside of the emergency department. This includes intensive care, critical care, coronary care, ambulatory care or acute medical admission units.
* Paramedics who are dual qualified and dual registered as another profession eg nurse- As this might influence data collection from the potential differences in prescriptive authority allowed from alternative professional registration.

Inclusion Criteria for Case Study Interview Participants:

- Participants must be an employee of the case study organisation and have relevant experience of PIP within the case study site. If required, informal discussions with potential participants expressing an interest will be used to confirm their eligibility and understanding of the research aims and objectives.

Exclusion Criteria for Case Study Interview Participants:

- No specific exclusion criteria will be set, however during recruitment, participants will be provided with written information about the study, to ensure they understand the research topic and aims, whilst ensuring they feel they are able to provide relevant data towards these through their participation in an interview.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Paramedics working in emergency departments and urgent care services who are qualified in independent prescribing and using this in their practice.
  2. Site staff employed at the case study sites who have experience and insights regarding paramedic prescribing in emergency and urgent care. These are anticipated to include senior and junior grade doctors, independent prescribing leads within the organisation, clinical managers, clinical directors and other healthcare professionals at the site, including nurses and non-prescribing paramedics.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Range and Frequency of Prescribed Medications | 6-8 months
  Demonstration of the range and frequency of prescribed medicines used by paramedic prescribers in different EUC settings, including cross case comparison to highlight if and how PIP is being used to contribute to patient care, if there are any limitations to PIP, alongside any differences between the different emergency and urgent care settings.
Understanding benefits and limitations of PIP | 6-8 months
  The development of a clear understanding of any benefits and limitations of PIP in these different EUC settings, including any contribution to patient care and healthcare service delivery, whilst also investigating any facilitators or barriers which influence this.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Latter, PhD, Study Chair — The University of Southampton
Locations (1):
- The University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
N/A- Participant data will not be shared